CLINICAL TRIAL: NCT01082159
Title: MiDAS II (Mild® Decompression Alternative to Open Surgery): Vertos Mild Patient Evaluation Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vertos Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MiDAS II
Record Dates: First submitted 2010-03-04; First posted 2010-03-08 (Estimated); Results first posted 2013-04-01 (Estimated); Last update posted 2013-04-01 (Estimated); Status verified 2013-02

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Spinal Stenosis; Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lumbar decompression (Other): Percutaneous lumbar decompression with mild® Device Kit.
  Interventions: Procedure: lumbar decompression

INTERVENTIONS:
Procedure: lumbar decompression — The mild® devices used in this study are specialized surgical instruments intended to be used to perform percutaneous lumbar decompressive procedures for the treatment of various spinal conditions.
  Other Names: The mild® Device Kit

SUMMARY:
This is a multi-center, prospective, patient outcomes assessment of Minimally Invasive Lumbar Decompression with the Mild® devices in patients with symptomatic central canal spinal stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic lumbar spinal stenosis (LSS) primarily caused by dorsal element hypertrophy.
* Prior failure of conservative therapy and Oswestry Disability Index (ODI) score > 20%.
* Radiologic evidence of lumbar spinal stenosis (LSS), ligamentum flavum hypertrophy (typically > 2.5 mm), confirmed by pre-op MRI and/or CT.
* Central canal cross sectional area clearly reduced per MRI/CT report.
* If present, anterior listhesis preferred ≤ 5.0mm and deemed stable by Investigator.
* Able to walk at least 10 feet unaided before being limited by pain.
* Available to complete 26 weeks of follow-up.
* A signed Informed Consent Form is obtained from the patient.
* Adults at least 18 years of age.

Exclusion Criteria:

* Prior surgery at intended treatment level.
* Compound fracture with interspinal retropulsion contributing to spinal stenosis.
* Disabling back or leg pain from causes other than LSS (e.g. acute compression fracture, metabolic neuropathy, or vascular claudication symptoms, etc.).
* Disc protrusion or osteophyte formation severe enough to confound study outcome.
* Facet hypertrophy severe enough to confound study outcome.
* Bleeding disorders and/or current use of anti-coagulants.
* Use of acetylsalicylic acid (ASA) and/or non-steroidal anti-inflammatory drug (NSAID) within 5 days of treatment.
* Epidural steroid administration within prior three weeks (of procedure).
* Inability of the patient to lie prone for any reason with anesthesia support (e.g.chronic obstructive pulmonary disease (COPD), obesity, etc.).
* Metabolic wound healing pathologies deemed by Investigator to compromise study outcomes.
* Dementia and/or inability to give informed consent.
* Pregnant and/or breastfeeding.
* On Workman's Compensation or considering litigation associated with back pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-02; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L Caraway, MD, PhD, Principal Investigator — The Center for Pain Relief Tri-State, PLLC; Bohdan W Chopko, MD, Principal Investigator — MedCentral Health System
Locations (8):
- United States (8):
  - Space Coast Pain Institute, Merritt Island, Florida
  - The Spine Center, Baltimore, Maryland
  - Occupational and Pain Management Professionals, Festus, Missouri
  - Lab2Marche, LLC, Las Vegas, Nevada
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - MedCentral Health System, Mansfield, Ohio
  - Kenneth Alo, MD, PA-TX, Houston, Texas
  - The Center for Pain Relief Tri-State, PLLC, Huntington, West Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from July 2008 through January 2010.
Groups:
- Lumbar Decompression: Single arm cohort having percutaneous decompression using the mild Device Kit
Period: Overall Study
Arm/Group | Lumbar Decompression
Started | 55
Completed | 46
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Lumbar Decompression
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 34
Age Continuous [Mean (Standard Deviation); unit: years] | 68.3 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Changes in Back Pain as Measured by a 10-point Visual Analog Scale (VAS).
Description: The 10-point Visual Analog Scale (VAS)rates 'no pain' as zero and 'worst pain imaginable' as ten. VAS mean improvement greater than or equal to 2 points is considered clinically relevant.
  The change from baseline to Month 6 is presented below where a positive value represents the baseline value minus the 6 month value.
Time Frame: Baseline and Month 6
Population: All available participants who reported Month 6 outcomes are included in this analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lumbar Decompression
Number analyzed (Participants) | 46
units on a scale | 3.59 [2.76 to 4.42]
Statistical Analysis 1: Comparison: Lumbar Decompression; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; change from baseline = 3.59, 95% CI 2-sided [2.76 to 4.42], Standard Deviation 2.87

2. Primary Outcome: Function as Measured Subjectively by the Oswestry Disability Index Questionnaire
Description: Oswestry Disability Index (ODI) measures permanent functional disability using questions regarding activities of daily living (ADL), specifically disturbance of ADL related to chronic back pain. Higher scores indicate a 'more limited' life. The ten topics of the ODI are rated from zero (no pain/limitation) to five (high pain/very limited physically). The worst possible score is 50 (100% disability) with the best score being zero (0% disability).Change from baseline to 6 months is presented below, where a positive value represents the baseline value minus the 6 month value.
Time Frame: Baseline and Month 6
Population: All available patients at 6 months are reported below.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Lumbar Decompression: Single arm cohort having percutaneous lumbar decompression using the mild Device Kit.
Arm/Group | Lumbar Decompression
Number analyzed (Participants) | 46
units on a scale | 12.17 [6.64 to 17.71]
Statistical Analysis 1: Comparison: Lumbar Decompression; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Change from Baseline = 12.17, 95% CI 2-sided [6.64 to 17.71], Standard Deviation 19.14

3. Primary Outcome: Quality of Life Changes as Determined by Short Form 12-question (SF-12) Survey Specifically Related to Physical Component Score (PCS).
Description: The SF-12 is a validated norm-based scoring tool used to determine treatment outcomes. The PCS summary measure shows the impact of the treatment on the patients abilities to conduct their usual physical activities. Clinical relevance of PCS is established by baseline to post-treatment improvement of 2 to 3 points. Norm-based scoring is used so that each scale has the same mean (50 points) and the same standard deviation (10 points) as the general US population in 1998. Scores below 50 indicate a decline in health status, with lower scores representing worse health status. Minimally Important Difference (MID) is a measure of true clinical relevance of a difference, with suggested MID for the Physical Component Summary (PCS) being 2 to 3 points. Change from baseline to 6 months is presented, where a positive value represents the 6 month value minus the baseline value.
Time Frame: Baseline and Month 6
Population: All participants at month 6 who completed all questionnaire fields necessary to analyze PCS data according to guidelines.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lumbar Decompression
Number analyzed (Participants) | 42
units on a scale | 8.32 [5.72 to 10.92]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of treatment through study period of six months.
Arm/Group | Lumbar Decompression
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less